CLINICAL TRIAL: NCT01704677
Title: Lumbar Disc Prosthesis Versus Multidisciplinary Rehabilitation in Chronic Back Pain and Localized Degenerative Disc. Long Term Follow-up of a Randomized Multicentre Trial
Brief Title: Lumbar Disc Prosthesis Versus Multidisciplinary Rehabilitation; 8-year Follow-up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: St. Olavs Hospital (Other); Haukeland University Hospital (Other); Helse Stavanger HF (Other Government); University Hospital of North Norway (Other)
Responsible Party: Principal Investigator, Kjersti Storheim, PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011/2177
Record Dates: First submitted 2012-10-02; First posted 2012-10-11 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Low Back Pain
Keywords: Chronic low back pain; Degenerated disc; Total disc replacement; Multidisciplinary rehabilitation; Long term results

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgery (Experimental): Replacement of the degenerative intervertebral lumbar disc with an artificial lumbar disc device (degeneration had to be restricted to the two lower levels (L4/L5 and/or L5/S1))
  Interventions: Procedure: Lumbar total disc replacement
- Multidiciplinary rehabilitation (Active Comparator)
  Interventions: Behavioral: Multidisciplinary rehabilitation

INTERVENTIONS:
Procedure: Lumbar total disc replacement — The surgical intervention consisted of replacement of the degenerative intervertebral lumbar disc with a artificial lumbar disc device in one or two of the lover lumbal levels (L4/L5 or/and L5/S1). The ProDisc consists of three pieces, two metal endplates and a polyethylene core that is fixed to the inferior endplate when the device is implanted, and is implanted through a retroperitoneal (or transperitoneal) access.
  Other Names: ProDisc II, Synthes Spine
  Arms: Surgery
Behavioral: Multidisciplinary rehabilitation — The intervention is based on a treatment model described by Brox et al (Spine 2003;28:1913-1921) and is also described in details by Hellum et al (BMJ, May 2011). It consisted of a cognitive approach and supervised physical exercise and was delivered by a team of physiotherapists and specialists in physical medicine and rehabilitation. The rehabilitation programme lasted for about 60 hours over three to five weeks.
  Arms: Multidiciplinary rehabilitation

SUMMARY:
During the past 25-30 years, surgery with total disc replacement (TDR) has become an option for a selection of patients with chronic low back pain (LBP) traditionally treated conservatively or operated on with spinal fusion. Randomized trials comparing TDR with fusion have found the clinical outcome of TDR at least equivalent to that of fusion, and the only study comparing TDR to non-surgical treatment (The Norwegian TDR study) concludes that TDR is significantly more effective than multidisciplinary rehabilitation (REHAB) after 2 years. However, the long-term effects of TDR in terms of clinical results, costs, reoperation- and revision rate, degenerative changes and prognostic factors have not been investigated in high quality prospective trials. This is very much required since TDR surgery is offered a great number of patients world wide, and is associated with high complexity and risk of serious complications and difficult revision. Hence, the overall aim of the present study is to evaluate the long term (eight years follow-up) effect of The Norwegian TDR study where TDR surgery were compared to modern multidisciplinary rehabilitation in patients with chronic low back pain and localized degenerative disc changes.

DETAILED DESCRIPTION:
Two-year results of the Norwegian TDR study were published in BMJ in May 2011 (Hellum et al). The current protocol is 8-year follow-up of patients included in the Norwegian TDR study.

Hypothesis of the 8-year follow-up:

Main hypothesis (H0): There are no differences in change between TDR and REHAB for pain and disability measured by Oswestry Disability Index (main outcome), back pain, quality of life, psychological variables, work status, patients satisfaction, drug use, urinary incontinence, and back surgeries after 8 years.

Secondary Hypothesis:

1. There are no differences in incidence and degree of disc degeneration at adjacent level or facet joint degeneration at index level between groups (radiological analysis).
2. There is no association between baseline characteristics, pelvic anatomy / sagittal balance (defined by lumbar lordosis, pelvic tilt, pelvic incidence angle and sacral slope), and clinical outcome after TDR.
3. There is no difference in cost effectiveness between surgery and REHAB 8 years after inclusion to the study.

Statistical analysis:

The investigators will use the same analysis as for 2-years results: two-way ANOVA, mixed model, regression analysis. p<0.05 will be considered statistically significant

Additional analysis (not conducted at 2 years):

1. cross-overs will receive last value before cross-over/fusion surgery
2. survival analysis
3. pelvic anatomy / sagittal balance (defined by lumbar lordosis, pelvic tilt, pelvic incidence angle and sacral slope) will be included in the predictor analysis
4. Both CT scans and MRI are taken for the evaluation of index level facet arthropathy

ELIGIBILITY:
Inclusion Criteria:

* aged 25-55 years
* had low back pain as the main symptom for at least 1 year
* structured physiotherapy or chiropractic treatment for at least 6 months without sufficient effect
* Oswestry Disability Index (ODI) of at least 30
* degenerative intervertebral disc changes in L4/L5 and/or L5/S1.Degeneration had to be restricted to the two lower levels. The following degenerative changes were evaluated: at least 40% reduction of disc height, Modic changes type I and/or II, high-intensity zone in the disc, and morphological changes classified as changes in signal intensity in the disc of grade 3 or 4. The disc was classified as degenerative if the first criteria alone or at least two changes were found on magnetic resonance imaging. The discs were independently classified by two observers (orthopaedic surgeon /radiologist). When in disagreement, the images were classified by a third observer and the outcome decided by simple majority.

Exclusion Criteria:

* Generalized chronic pain syndrome (widespread myofascial pain)
* Degeneration established in more than two levels. To be classified as a normal disc, the disc height must not be reduced more than 40% and all other criteria of degenerative disc disease aforementioned must be absent. The classification of a normal disc is performed by two independent observers. If disagreement, the pictures will be classified by a third observer and the outcome decided by simple majority.
* Symptoms of spinal stenosis
* Disc protrusion or recess stenosis with nerve root affection
* Spondylolysis
* Isthmic spondylolisthesis
* Arthritis
* Former fracture of L1 - S1
* Ongoing psychiatric or somatic disease that excludes either one or both treatment alternatives
* Does not understand Norwegian language, spoken or in writing
* Drug abuse
* Osteoporosis
* Congenital or acquired deformity

Patients were examined by an orthopaedic surgeon and a specialist in physical medicine and rehabilitation together, which had to agree on inclusion.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 151 (Actual)
Dates: Start 2012-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index Oswestry Disability Index | Baseline, 6 weeks, 3 months, 6 months, 1, 2 and 8 years after inclusion to trial
  Version 2.0

SECONDARY OUTCOMES:
Low back pain | Baseline, 6 weeks, 3 months, 6 months, 1, 2 and 8 years after inclusion to trial
  Measured by a VAS scale (0-100 mm)
EQ-5D | Baseline, 6 weeks, 3 months, 6 months, 1, 2 and 8 years after inclusion to trial
  general health status
HSCL-25 | Baseline, 3 months, 6 months, 1, 2 and 8 years after inclusion to trial
  Hopkins Symptom Check List 25 for emotional distress
Work status | Baseline, 6 weeks, 3 months, 6 months, 1, 2 and 8 years after inclusion to trial
Satisfaction with treatment outcome | Baseline, 6 weeks, 3 months, 6 months, 1, 2 and 8 years after inclusion to trial
  7 point Likert scale
Satisfaction with care | Baseline, 6 weeks, 3 months, 6 months, 1 and 8 years after inclusion to trial
  5 point Likert scale
Drug consumption | Baseline, 6 weeks, 3 months, 6 months, 1, 2 and 8 years after inclusion to trial
  Daily, weekly, type
Urinary incontinence | Baseline, 3 months, 6 months, 1, 2 and 8 years after inclusion to trial
  Stress incontinence, urge incontinence
Back surgeries and multidisciplinary rehabilitation | Baseline, 6 weeks, 3 months, 6 months, 1, 2 and 8 years after inclusion to trial
  All surgeries and multidisciplinary rehabilitation due to low back pain will be registered
Disc degeneration | Baseline, 2 and 8 years after inclusion to trial
  Disc degeneration at adjacent level
Facet joint degeneration | Baseline, 2 and 8 years after inclusion to trial
  Facet joint degeneration at index level
Cost-effectiveness | Baseline, 6 weeks, 3 months, 6 months, 1, 2 and 8 years after inclusion to trial
  The EQ-5D questionnaire will be used to estimate patient utilities

OTHER OUTCOMES:
Time to surgery | From baseline to 8 years after inclusion to the study
  For patients randomized to TDR surgery: time to fixation
  For patients randomized to REHAB: time to TDR surgery or fixation

CONTACTS AND LOCATIONS:
Overall Officials: Kjersti Storheim, PhD, Principal Investigator — Oslo University Hospital Ullevål
Locations (1):
- Oslo University Hospital Ullevål, Oslo, Oslo County, Norway

REFERENCES:
- [Background] Hellum C, Johnsen LG, Storheim K, Nygaard OP, Brox JI, Rossvoll I, Ro M, Sandvik L, Grundnes O; Norwegian Spine Study Group. Surgery with disc prosthesis versus rehabilitation in patients with low back pain and degenerative disc: two year follow-up of randomised study. BMJ. 2011 May 19;342:d2786. doi: 10.1136/bmj.d2786. PMID 21596740
- [Background] Hellum C, Johnsen LG, Gjertsen O, Berg L, Neckelmann G, Grundnes O, Rossvoll I, Skouen JS, Brox JI, Storheim K; Norwegian Spine Study Group. Predictors of outcome after surgery with disc prosthesis and rehabilitation in patients with chronic low back pain and degenerative disc: 2-year follow-up. Eur Spine J. 2012 Apr;21(4):681-90. doi: 10.1007/s00586-011-2145-3. Epub 2012 Jan 13. PMID 22246644
- [Background] Hellum C, Berg L, Gjertsen O, Johnsen LG, Neckelmann G, Storheim K, Keller A, Grundnes O, Espeland A; Norwegian Spine Study Group. Adjacent level degeneration and facet arthropathy after disc prosthesis surgery or rehabilitation in patients with chronic low back pain and degenerative disc: second report of a randomized study. Spine (Phila Pa 1976). 2012 Dec 1;37(25):2063-73. doi: 10.1097/BRS.0b013e318263cc46. PMID 22706091
- [Background] Johnsen LG, Hellum C, Storheim K, Nygaard OP, Brox JI, Rossvoll I, Ro M, Andresen H, Lydersen S, Grundnes O, Pedersen M, Leivseth G, Olafsson G, Borgstrom F, Fritzell P; Norwegian Spine Study Group. Cost-effectiveness of total disc replacement versus multidisciplinary rehabilitation in patients with chronic low back pain: a Norwegian multicenter RCT. Spine (Phila Pa 1976). 2014 Jan 1;39(1):23-32. doi: 10.1097/BRS.0000000000000065. PMID 24150435
- [Background] Berg L, Hellum C, Gjertsen O, Neckelmann G, Johnsen LG, Storheim K, Brox JI, Eide GE, Espeland A; Norwegian Spine Study Group. Do more MRI findings imply worse disability or more intense low back pain? A cross-sectional study of candidates for lumbar disc prosthesis. Skeletal Radiol. 2013 Nov;42(11):1593-602. doi: 10.1007/s00256-013-1700-x. Epub 2013 Aug 28. PMID 23982421
- [Background] Johnsen LG, Hellum C, Nygaard OP, Storheim K, Brox JI, Rossvoll I, Leivseth G, Grotle M. Comparison of the SF6D, the EQ5D, and the oswestry disability index in patients with chronic low back pain and degenerative disc disease. BMC Musculoskelet Disord. 2013 Apr 26;14:148. doi: 10.1186/1471-2474-14-148. PMID 23622053
- [Background] Johnsen LG, Brinckmann P, Hellum C, Rossvoll I, Leivseth G. Segmental mobility, disc height and patient-reported outcomes after surgery for degenerative disc disease: a prospective randomised trial comparing disc replacement and multidisciplinary rehabilitation. Bone Joint J. 2013 Jan;95-B(1):81-9. doi: 10.1302/0301-620X.95B1.29829. PMID 23307678
- [Background] Berg L, Gjertsen O, Hellum C, Neckelmann G, Johnsen LG, Eide GE, Espeland A. Reliability of change in lumbar MRI findings over time in patients with and without disc prosthesis--comparing two different image evaluation methods. Skeletal Radiol. 2012 Dec;41(12):1547-57. doi: 10.1007/s00256-012-1394-5. Epub 2012 Mar 20. PMID 22430564
- [Derived] Garratt AM, Furunes H, Hellum C, Solberg T, Brox JI, Storheim K, Johnsen LG. Evaluation of the EQ-5D-3L and 5L versions in low back pain patients. Health Qual Life Outcomes. 2021 May 28;19(1):155. doi: 10.1186/s12955-021-01792-y. PMID 34049574